CLINICAL TRIAL: NCT04474743
Title: Multi-center, Controlled Cross-sectional Analysis of the Phenotype of Malnutrition in Patients With Liver Cirrhosis, Chronic Pancreatitis and Short Bowel Syndrome (as Part of the Joint Project "Enteral Nutrition in Malnutrition Due to Diseases of the Gastrointestinal Tract: From Basic Understanding to an Innovative Treatment Concept" (EnErGie))
Brief Title: Malnutrition in Chronic Gastrointestinal Diseases, Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: University Medical Center Rostock (Other); University of Applied Sciences Neubrandenburg (Other); Leibniz Institute for Farm Animal Biology (FBN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: A 2018-0129
Record Dates: First submitted 2020-06-29; First posted 2020-07-17 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Liver Cirrhoses; Chronic Pancreatitis; Short Bowel Syndrome
MeSH Terms: conditions — Pancreatitis, Chronic; Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Plasma, Faeces, Urine, Proximal Small Intestinal Biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Liver Cirrhosis: Patients diagnosed with liver cirrhosis.
  Interventions: Other: No intervention - cross-sectional observational only
- Chronic Pancreatitis: Patients diagnosed with chronic pancreatitis.
  Interventions: Other: No intervention - cross-sectional observational only
- Short Bowel Syndrome: Patients diagnosed with short bowel Syndrome.
  Interventions: Other: No intervention - cross-sectional observational only
- Control Patients: Otherwise healthy patients visiting hospital with other non-severe diseases.
  Interventions: Other: No intervention - cross-sectional observational only
- Healthy Controls: Healthy subjects recruited from the general population.
  Interventions: Other: No intervention - cross-sectional observational only

INTERVENTIONS:
Other: No intervention - cross-sectional observational only — No intervention - cross-sectional observational only

SUMMARY:
Malnutrition and muscle wasting are common consequences of life-threatening, chronic diseases of the gastrointestinal tract. Such diseases include liver cirrhosis, chronic pancreatitis and short bowel syndrome. Malnutrition and muscle wasting increase the risk of complications, reduce the life expectancy and impair the quality of life. The development of malnutrition and muscle wasting is different, as is the diagnosis and nutritional treatment. There are also different mechanisms of origin for the underlying diseases. The aim of the study is to compare data related to nutrition and physical condition of patients with liver cirrhosis, chronic pancreatitis and short bowel syndrome. Malnutrition and muscle wasting within the specific diseases will be characterized and possible correlations will be identified.

For this, malnourished and non-malnourished patients of the different diseases are compared with controls patients with non-specific complaints of the gastrointestinal tract as well as with healthy study participants.

Data on food intake, physical activity, body composition and body measurements as well as muscle strength and muscle function are recorded. Blood values as well as transport and barrier properties of the intestine will also be examined.

DETAILED DESCRIPTION:
Malnutrition and sarcopenia are consequences of life-threatening gastroenterological diseases such as liver cirrhosis, chronic pancreatitis and short bowel syndrome and are associated with a poorer clinical outcome and a reduced quality of life. The diagnostic criteria of both conditions differ, as do the consequences for adequate nutritional therapy. Nevertheless, malnutrition and sarcopenia are often discussed in confusion in the literature. In addition, the underlying mechanisms of malnutrition and sarcopenia can differ in the various diseases. The aim of the study is to compare nutrition-associated parameters from patients with liver cirrhosis, chronic pancreatitis and short bowel syndrome, to characterize the disease-specific phenotype of malnutrition and sarcopenia of the examined diseases and to obtain information on mechanistic relationships. The pathophysiological understanding of the clinical settings as well as the development of malnutrition and sarcopenia is important for choosing specific nutritional therapies. For this, malnourished and non-malnourished patients of each examined disease are compared with controls from patients with non-specific, abdominal symptoms and healthy control subjects. Data on food intake, physical activity, body composition and anthropometry as well as muscle strength and muscle function are recorded. Clinical and chemical blood parameters, the plasma metabolome as well as transport and barrier proteins of the intestine are also examined.

ELIGIBILITY:
Inclusion Criteria:

Liver Cirrhosis:

* based on clinical and imaging criteria (sonography or computed tomography (CT) or magnetic resonance imaging (MRI)) without evidence of hepatocellular carcinoma
* Child-Pugh Stadium A-C

Chronic Pancreatitis:

* based on imaging criteria (endoscopic ultrasound, computed tomography (CT), magnetic resonance imaging (MRI), magnetic resonance cholangiopancreatography (MRCP))
* large and small duct disease
* with or without exocrine insufficiency
* with or without endocrine insufficiency
* patients after left pancreatic resection or pancreaticojejunostomy or duodenal pancreatic head resection

Short Bowel Syndrome (SBS):

- based on clinical anamnestic criteria and state after bowel resection followed by primary or secondary oral autonomy (intestinal failure)

Control Patients:

* patients without known underlying gastroenterological disease with an indication for esophago-gastro-duodenoscopy for symptom clarification
* negative Nutritional Risk Screening (NRS-2002 < 3)
* gastroscopy without clinically relevant result (mild gastritis aspect, small axial hernia, typical glandular cysts, typical brunneromas can be included)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

General Exclusion Criteria:

* parenteral nutrition in the previous 6 months
* pacemaker or implanted defibrillator
* pregnancy or lactation
* lack of ability to answer the questionnaires
* taking certain medications during the previous 4 weeks (protein pump inhibitors and H2 antagonists, except medication on demand or ≤ 4 weeks continuously, antibiotics, narcotics, non-opioid analgesics except medication on demand (≤ 1 day/week), anticholinergics, antidepressants, motility drugs (metoclopramide, motilium, bromocriptine, prucalopride), thyroid drugs except stable thyroid hormone substitution with euthyroid metabolism, steroids, immunomodulators, anti-inflammatory biologics)

Subsequent Exclusion of Control Patients:

* if, contrary to expectations, malnutrition is diagnosed in spite of an inconspicuous NRS-2002 within the framework of the study
* as well as in the case of relevant, conspicuous esophago-gastro-duodenoscopy findings

Specific Exclusion Criteria:

Liver Cirrhosis:

* steatohepatitis according to clinical or laboratory parameters
* acute alcoholic hepatitis according to clinical and imaging parameters (sonography, CT, MRI)
* existing transjugular intrahepatic portosystemic shunt (TIPS)
* known hepatocellular carcinoma (HCC)
* state after liver transplantation

Chronic Pancreatitis:

* acute pancreatitis
* extrapancreatic infection
* coexisting liver cirrhosis based on clinical and imaging parameters
* state after surgery with alteration of food flow (partial or total pancreaticoduodenectomy)
* known pancreatic carcinoma or state after therapy of pancreatic carcinoma (surgery or chemotherapy or radiation)

Short Bowel Syndrome (SBS):

* acute phase of intestinal insufficiency (less than 28 days after resection)
* intravenous substitution of macronutrients (water, electrolytes, glucose, amino acids or lipids (intestinal insufficiency)
* intramuscular substitution of micronutrients is allowed (e.g. vitamin B12)
* uncontrolled underlying disease leading to SBS (e.g. active Crohn's disease)

Control Patients:

* major underlying and concomitant diseases
* food allergies

Healthy controls:

* tumor diseases in the past 5 years
* medically diagnosed, serious chronic diseases or changes in the gastrointestinal tract that may affect the absorption of nutrients (e.g. celiac disease, chronic inflammatory bowel disease or irritable bowel syndrome diagnosed according to Rome IV criteria, relevant bowel resections including short bowel syndrome)
* rheumatic diseases requiring permanent drug therapy (rheumatoid arthritis, fibromyalgia)
* chronic use of anti-inflammatory or pain-relieving drugs or use of anti-inflammatory or pain-relieving drugs for more than 3 days in the last 3 weeks
* average daily alcohol consumption > 20 g in women and > 30 g in men
* diagnosed severe liver disease requiring medical attention and drug therapy (liver cirrhosis, non-alcoholic steatohepatitis (NASH) / alcoholic steatohepatitis (ASH), hepatitides)
* acute or chronic pancreatitis
* acute and chronic renal failure
* myocardial infarction or cerebral insult within 6 months prior to examination
* coronary artery disease/pAVK (peripheral artery disease (PAD))
* heart failure with stages 3 and 4 according to NYHA (New York Heart Association) classification
* severe chronic pulmonary disease (COPD)
* history of significant neurological or psychiatric diseases (including epilepsy, bipolar disorders, dementia and neuromuscular diseases)
* presence of pareses including mono- and diparesis
* rare congenital metabolic diseases (cystic fibrosis, phenylketonuria)
* expected altered body composition (extreme sports activity < 2h/day), edema, amputation of the extremities (arm and/or leg)
* highly atypical or restrictive dietary choices/concepts followed voluntarily (macrobiotics, paleo-diet, Atkins diet, Mayo diet, instinctive diets) or due to food intolerances/allergies
* simultaneous participation in other studies associated with drug use and potentially having a significant impact on body composition or dietary behaviour

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients eligible for study participation will be recruited at the University hospitals in the cities of Rostock and Greifswald (Northeast Germany). Hospitalized as well outcare-patients will be considered for recruitment. Healthy controls will be recruited from the general public in the city of Neubrandenburg (Northeast Germany).
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Sarcopenia | Baseline
  Descriptive and inferential determination of the prevalence of sarcopenia according to the European Working Group on Sarcopenia in Older People 2 criteria (EWGSOP2 criteria) in malnourished and non malnourished patients with liver cirrhosis, chronic pancreatitis or short bowel syndrome - as a total group and separated by type of disease
Quantitative Food Intake | Baseline
  Determination of quantitative food intake assessed by the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Qualitative Food Intake | Baseline
  Determination of qualitative food intake assessed by the Study of Health in Pomerania Food Frequency Questionnaire (SHIP-FFQ) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Physical Activity | Baseline
  Determination of physical activity assessed by the International Physical Activity Questionnaire (IPAQ) Short Form in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Body Weight | Baseline
  Determination of body weight measured in kilograms in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Height | Baseline
  Determination of height measured in meters in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Body Mass Index | Baseline
  Determination of body mass index in kg/m^2 (calculated from the values obtained for body weight and height) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Waist Circumference | Baseline
  Determination of waist circumference measured in centimeters in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Hip Circumference | Baseline
  Determination of hip circumference measured in centimeters in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Waist-to-Hip Ratio | Baseline
  Determination of waist-to-hip ratio (calculated from the values obtained for waist and hip circumference) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Upper Arm Circumference | Baseline
  Determination of upper arm circumference measured in centimeters in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Triceps Skinfold Thickness | Baseline
  Determination of triceps skinfold thickness measured in millimeters in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Fat Free Mass | Baseline
  Determination of fat free mass measured by Bioelectrical Impedance Analysis (BIA) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Skeletal Muscle Mass | Baseline
  Determination of skeletal muscle mass measured by Bioelectrical Impedance Analysis (BIA) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Fat Mass | Baseline
  Determination of fat mass measured by Bioelectrical Impedance Analysis (BIA) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Total Body Water | Baseline
  Determination of total body water measured by Bioelectrical Impedance Analysis (BIA) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Extracellular Water | Baseline
  Determination of extracellular water measured by Bioelectrical Impedance Analysis (BIA) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Phase Angle | Baseline
  Determination of phase angle measured by Bioelectrical Impedance Analysis (BIA) in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Muscle Strength | Baseline
  Determination of muscle strength measured by a handgrip strength dynamometer in comparison with non malnourished and non-sarcopenia patients and in comparison with healthy control subjects
Hemoglobin | Baseline
  Determination of hemoglobin level in comparison to control patients and in comparison to healthy control subjects
Hematocrit | Baseline
  Determination of hematocrit level in comparison to control patients and in comparison to healthy control subjects
Mean Corpuscular Volume | Baseline
  Determination of mean corpuscular volume in comparison to control patients and in comparison to healthy control subjects
Mean Corpuscular Hemoglobin Concentration | Baseline
  Determination of mean corpuscular hemoglobin concentration in comparison to control patients and in comparison to healthy control subjects
Reticulocyte Count | Baseline
  Determination of reticulocyte count in comparison to control patients and in comparison to healthy control subjects
Sodium | Baseline
  Determination of plasma concentration of sodium in comparison to control patients and in comparison to healthy control subjects
Potassium | Baseline
  Determination of plasma concentration of potassium in comparison to control patients and in comparison to healthy control subjects
Calcium | Baseline
  Determination of plasma concentration of calcium in comparison to control patients and in comparison to healthy control subjects
Magnesium | Baseline
  Determination of plasma concentration of magnesium in comparison to control patients and in comparison to healthy control subjects
Phosphate | Baseline
  Determination of plasma concentration of phosphate in comparison to control patients and in comparison to healthy control subjects
Aspartate Transaminase | Baseline
  Determination of plasma concentration of aspartate transferase in comparison to control patients and in comparison to healthy control subjects
Alanine Aminotransferase | Baseline
  Determination of plasma concentration of alanine aminotransferase in comparison to control patients and in comparison to healthy control subjects
Gamma-glutamyl Transferase | Baseline
  Determination of plasma concentration of gamma-glutamyl transferase in comparison to control patients and in comparison to healthy control subjects
Alkaline Phosphatase | Baseline
  Determination of plasma concentration of alkaline phosphatase in comparison to control patients and in comparison to healthy control subjects
Bilirubin | Baseline
  Determination of plasma concentration of bilirubin in comparison to control patients and in comparison to healthy control subjects
C-reactive Protein | Baseline
  Determination of plasma concentration of C-reactive protein in comparison to control patients and in comparison to healthy control subjects
Interleukin-1 Beta | Baseline
  Determination of serum concentration of interleukin-1 beta in comparison to control patients and in comparison to healthy control subjects
Interleukin-6 | Baseline
  Determination of plasma concentration of interleukin-6 in comparison to control patients and in comparison to healthy control subjects
Tumor Necrosis Factor Alpha | Baseline
  Determination of serum concentration of tumor necrosis factor alpha in comparison to control patients and in comparison to healthy control subjects
Albumin | Baseline
  Determination of plasma concentration of albumin in comparison to control patients and in comparison to healthy control subjects
Creatinine | Baseline
  Determination of plasma concentration of creatinine in comparison to control patients and in comparison to healthy control subjects
Urea | Baseline
  Determination of plasma concentration of urea in comparison to control patients and in comparison to healthy control subjects
Uric Acid | Baseline
  Determination of plasma concentration of uric acid in comparison to control patients and in comparison to healthy control subjects
Glucose | Baseline
  Determination of plasma concentration of glucose in comparison to control patients and in comparison to healthy control subjects
Glycated hemoglobin | Baseline
  Determination of plasma concentration of glycated hemoglobin in comparison to control patients and in comparison to healthy control subjects
Insulin | Baseline
  Determination of plasma concentration of insulin in comparison to control patients and in comparison to healthy control subjects
Total Cholesterol | Baseline
  Determination of plasma concentration of total cholesterol in comparison to control patients and in comparison to healthy control subjects
High-density Lipoprotein Cholesterol | Baseline
  Determination of plasma concentration of high-density lipoprotein cholesterol in comparison to control patients and in comparison to healthy control subjects
Low-density Lipoprotein Cholesterol | Baseline
  Determination of plasma concentration of low-density lipoprotein cholesterol in comparison to control patients and in comparison to healthy control subjects
Triglycerides | Baseline
  Determination of plasma concentration of triglycerides in comparison to control patients and in comparison to healthy control subjects
Non-essential Fatty Acids | Baseline
  Determination of plasma concentration of non-essential fatty acids in comparison to control patients and in comparison to healthy control subjects
Zinc | Baseline
  Determination of serum concentration of zinc in comparison to control patients and in comparison to healthy control subjects
Iron | Baseline
  Determination of plasma concentration of iron in comparison to control patients and in comparison to healthy control subjects
Plasma Metabolome | Baseline
  In a participants subgroup, investigations of the plasma metabolome in comparison with control patients and in comparison with healthy control subjects
Intestinal Barrier Function | Baseline
  Determination of the intestinal barrier function in a patient subgroup in comparison to control patients (using proximal small intestinal biopsies, qRT-PCR (Real Time Polymerase Chain Reaction) of different intestinal barrier markers)
Expression of Intestinal Ion Transporters | Baseline
  Determination of the expression of intestinal ion transporters in a patient subgroup in comparison to control patients (using proximal small intestinal biopsies, qRT-PCR (Real Time Polymerase Chain Reaction) of different intestinal transport markers)

SECONDARY OUTCOMES:
Malnutrition-Sarcopenia Score | Baseline
  Correlative, factorial or other presentation of the results including statistical-mathematical argumentation of the usefulness of a combined malnutrition-sarcopenia score (MaSa score) for practical application.
Validity of the Study of Health in Pomerania Food Frequency Questionnaire | Baseline
  Determination of the validity of the Study of Health in Pomerania Food Frequency Questionnaire (SHIP-FFQ) by assessment of percent agreement with the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ)
Factor Analysis of Phenotypes of Sarcopenia and Malnutrition | Baseline
  Determination of parameters characterizing phenotypes of sarcopenia and malnutrition in the investigated gastroenterological disease (liver cirrhosis, chronic pancreatitis, short bowel syndrome) by factor analysis

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Lamprecht, Principal Investigator — University Medicine Rostock
Locations (3):
- Germany (3):
  - University Medicine Greifswald, Greifswald
  - University of Applied Sciences Neubrandenburg, Neubrandenburg
  - Univeristy Medicine Rostock, Rostock

REFERENCES:
- [Derived] Wiese ML, Gartner S, von Essen N, Doller J, Frost F, Tran QT, Weiss FU, Meyer F, Valentini L, Garbe LA, Metges CC, Bannert K, Sautter LF, Ehlers L, Jaster R, Lamprecht G, Steveling A, Lerch MM, Aghdassi AA. Malnutrition Is Highly Prevalent in Patients With Chronic Pancreatitis and Characterized by Loss of Skeletal Muscle Mass but Absence of Impaired Physical Function. Front Nutr. 2022 Jun 1;9:889489. doi: 10.3389/fnut.2022.889489. eCollection 2022. PMID 35719155